CLINICAL TRIAL: NCT00655681
Title: Prevention of Post Operative Bone Loss in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 07-213
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Results first posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-07

CONDITIONS: Osteoporosis; Cerebral Palsy; Spina Bifida; Osteopenia; Osteogenesis Imperfecta
Keywords: pediatric osteoporosis; pediatric osteopenia; pamidronate; post operative osteopenia
MeSH Terms: conditions — Osteoporosis; Cerebral Palsy; Spinal Dysraphism; Bone Diseases, Metabolic; Osteogenesis Imperfecta; Juvenile osteoporosis | interventions — Pamidronate; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A recieveds pamidronate 1mg/kg once (Experimental): Receives pamidronate 1mg/kg once
  Interventions: Drug: pamidronate
- B: placebo group recieves saline (Placebo Comparator): receives saline injection 10 cc/kg over 4 hours once post operatively
  Interventions: Other: saline

INTERVENTIONS:
Drug: pamidronate — The pamidronate is mixed 1 to 10 (10 cc of saline for each 1 mg pamidronate), with a minimum volume of 50 cc saline. The medication is administered as an IV infusion to run at a rate beginning at 20 cc/hr, adjusting the rate so that the infusion will run over 4 hours. For children < 8 kg (80cc infusion), the rate would be 20 cc/hr and the duration would be determined by the volume.
  Other Names: Aredia
  Arms: A recieveds pamidronate 1mg/kg once
Other: saline — receives saline 10cc/kg over 4 hours post operatively in addition to routine post operative fluids
  Other Names: normal saline
  Arms: B: placebo group recieves saline

SUMMARY:
Hypothesis: one-dose pamidronate will prevent post-operative bone loss in children at risk for low bone density

Plan: children with chronic disease such as CP, spina bifida, etc. will be recruited pre operatively and studied with DXA scan. After surgery, children will be randomized to receive either pamidronate or saline. Repeat DXA scan will determine bone lost after end of immobilization or nonweightbearing.

DETAILED DESCRIPTION:
Children at risk for post operative bone loss will be studied with preoperative DXA scan of spine and distal femora

Preoperative screening with standard labs electrolytes, Ca++, PO4, creatinine, Vit D

Following surgery of hip(s) or lower extremities, randomization into treatment with low dose IV pamidronate (one dose) v placebo group

Repeat DXA scan after end of immobilization or non-weightbearing

ELIGIBILITY:
Inclusion Criteria:

* chronic condition predisposing to low bone density, such as cerebral palsy, osteogenesis imperfecta
* lower extremity surgery proposed that will require post op nonweightbearing, casted or not, for a minimum of 4 weeks

Exclusion Criteria:

* creatinine >1.2
* prior bisphosphonate exposure
* orthopaedic implants in distal femoral precluding DXA scan
* inability to cooperate with DXA scan

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2007-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Szalay, MD, Principal Investigator — University of New Mexico Carrie Tingley Hospital
Locations (1):
- University of New Mexico Carrie Tingley Hospital, Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 2007 and 2011, twenty-four subjects were enrolled, and 20 were included in the final analysis (2 subjects were not administered drug due to slightly low serum calcium, and two did not return for the final dual energy x-ray absorptiometry (DXA) scan). There were 11 subjects randomized into the treatment group and 9 into the control group.
Pre-assignment Details: 2 subjects were not administered drug due to slightly low serum calcium, and two did not return for the final DXA scan
Groups:
- A Patients Receiving Pamidronate: Receives pamidronate 1mg/kg IV once during the post operative period. Pamidronate is given over 4 hours.
- B Patients Receiving Saline (Control Placebo): receives saline injection IV once in the post operative period in addition to routine post operative fluids.
Period: Overall Study
Arm/Group | A Patients Receiving Pamidronate | B Patients Receiving Saline (Control Placebo)
Started | 12 | 10
Completed | 11 (Did not return for final DXA) | 9
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: Children at risk for low bone density who were to undergo orthopaedic surgical procedure that would result in cast immobilization or non weight bearing for at least 4 weeks
Groups:
- A: Recieved Pamidronate 1mg/kg: Receives pamidronate 1mg/kg IV once. The pamidronate is mixed 1 to 10 (10 cc of saline for each 1 mg pamidronate), with a minimum volume of 50 cc saline. The medication is administered as an IV infusion to run at a rate beginning at 20 cc/hr, adjusting the rate so that the infusion will run over 4 hours. For children < 8 kg (80cc infusion), the rate would be 20 cc/hr and the duration would be determined by the volume.
- B: Receives Saline 10cc/kg: receives saline injection IV once 10cc/kg over 4 hours post operatively in addition to routine post operative fluids
- Total: Total of all reporting groups
Arm/Group | A: Recieved Pamidronate 1mg/kg | B: Receives Saline 10cc/kg | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Continuous [Mean (Full Range); unit: years] | 9.1 [4 to 14] | 7.8 [4 to 12] | 8.5 [4 to 14]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 9 | 20
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 7 | 1 | 8
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Amount of Bone Density Lost (%) From pre-to Post-operative DXA Scan
Description: Mean change lumbar spine post-op BMD Mean Right metaphyseal femur change post op BMD Mean Right transitional femur change post op BMD Mean Right diaphyseal femur change post op BMD
  Mean Left metaphyseal femur change post op BMD Mean Left transitional femur change post op BMD Mean Left diaphyseal femur change post op BMD
Time Frame: Preoperative to post-operative DXA scan (4-12 weeks)
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- A Patients Receiving Pamidronate: Receives pamidronate 1mg/kg one time post operatively over 4 hours
- B Patients Receiving Saline (Control Placebo): receives saline injection once 10 cc/kg over 4 hours in additional to routine post op fluide
Arm/Group | A Patients Receiving Pamidronate | B Patients Receiving Saline (Control Placebo)
Number analyzed (Participants) | 11 | 9
percent change | 0.043 (0.04) | -0.025 (0.02)

ADVERSE EVENTS:
Time Frame: no adverse event encountered in 4 years
Groups:
- A: Receives Pamidronate 1mg/kg: Receives pamidronate 1mg/kg : The pamidronate is mixed 1 to 10 (10 cc of saline for each 1 mg pamidronate), with a minimum volume of 50 cc saline. The medication is administered as an IV infusion to run at a rate beginning at 20 cc/hr, adjusting the rate so that the infusion will run over 4 hours. For children < 8 kg (80cc infusion), the rate would be 20 cc/hr and the duration would be determined by the volume.
- B: Receives Saline 10cc/kg Over 4 Hours Post Operatively: receives saline injection: receives saline 10cc/kg over 4 hours post operatively in addition to routine post operative fluids
Arm/Group | A: Receives Pamidronate 1mg/kg | B: Receives Saline 10cc/kg Over 4 Hours Post Operatively
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 0/11 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No